CLINICAL TRIAL: NCT00416455
Title: Utility of Preoperative FDG-PET/CT Scanning Prior to Primary Chemoradiation Therapy to Detect Retroperitoneal Lymph Node Metastasis in Patients With Locoregionally Advanced Carcinoma of the Cervix (IB2, IIA ≥ 4 CM, IIB-IVA) or Endometrium (Grade 3 Endometrioid Endometrial Carcinoma; Serous Papillary Carcinoma, Clear Cell Carcinoma, or Carcinosarcoma (Any Grade); and Grade 1 OR 2 Endometrioid Endometrial Carcinoma With Cervical Stromal Involvement Overt in Clinical Examination or Confirmed by Endocervical Curettage
Brief Title: Fludeoxyglucose (FDG) F 18 PET Scan, CT Scan, and Ferumoxtran-10 MRI Scan Before Chemotherapy and Radiation Therapy in Finding Lymph Node Metastasis in Patients With Locally Advanced Cervical Cancer or High-Risk Endometrial Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NCI-2009-00600; NCI-2009-00600 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000521453; ACRIN 6671; GOG-0233/ACRIN 6671; GOG-0233-ACRIN 6671 (Other: NRG Oncology); GOG-0233 (Other: CTEP); U10CA180868 (NIH); U10CA027469 (NIH)
Record Dates: First submitted 2006-12-27; First posted 2006-12-28 (Estimated); Results first posted 2015-12-14 (Estimated); Last update posted 2019-07-23 (Actual); Status verified 2018-11

CONDITIONS: Cervical Adenocarcinoma; Cervical Adenosquamous Cell Carcinoma; Cervical Small Cell Carcinoma; Cervical Squamous Cell Carcinoma; Endometrial Clear Cell Carcinoma; Endometrial Papillary Serous Carcinoma; Stage I Endometrial Carcinoma; Stage IB Cervical Cancer; Stage II Endometrial Carcinoma; Stage IIA Cervical Cancer; Stage IIB Cervical Cancer; Stage III Cervical Cancer; Stage III Endometrial Carcinoma; Stage IVA Cervical Cancer
MeSH Terms: conditions — Endometrial Neoplasms; Uterine Cervical Neoplasms | interventions — Fluorodeoxyglucose F18; Magnetic Resonance Spectroscopy; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole; ferumoxtran-10; Sentinel Lymph Node Biopsy

ARMS (1):
- Treatment (diagnostic scans, surgery, chemotherapy, radiation) (Experimental): Patients receive fludeoxyglucose F 18 (FDG) IV followed 60 minutes later by positron emission tomography (PET)/CT scanning on day 1. Patients also receive ferumoxtran-10 IV over 30-45 minutes on day 1 (or 24-36 hours before MRI) and undergo MRI on day 2. Patients undergo extraperitoneal, laparoscopic, or trans-peritoneal lymphadenectomy with pelvic and abdominal lymph node biopsy within 2 weeks after PET/CT scan. Patients diagnosed with metastatic disease prior to lymph node biopsy proceed directly to primary treatment. Patients with cervical cancer undergo chemoradiotherapy within 4 weeks of PET/CT scan.
  Interventions: Radiation: fludeoxyglucose F 18; Procedure: positron emission tomography; Procedure: computed tomography; Drug: ferumoxtran-10; Procedure: magnetic resonance imaging; Procedure: diagnostic lymphadenectomy; Procedure: lymph node biopsy

INTERVENTIONS:
Radiation: fludeoxyglucose F 18 — Undergo FDG PET/CT
  Other Names: 18FDG; FDG
Procedure: positron emission tomography — Undergo FDG PET/CT
  Other Names: FDG-PET; PET; PET scan; tomography, emission computed
Procedure: computed tomography — Undergo FDG PET/CT
  Other Names: tomography, computed
Drug: ferumoxtran-10 — Undergo femoxtran-10 MRI
  Other Names: AMI-227; Combidex; G-53425; Sinerem; USPIO
Procedure: magnetic resonance imaging — Undergo femoxtran-10 MRI
  Other Names: MRI; NMR imaging; NMRI; nuclear magnetic resonance imaging
Procedure: diagnostic lymphadenectomy — Undergo extraperitoneal, laparoscopic, or trans-peritoneal lymphadenectomy
Procedure: lymph node biopsy — Undergo pelvic and abdominal lymph node biopsy
  Other Names: Biopsy of Lymph Node

SUMMARY:
This phase I/II trial is studying how well fludeoxyglucose F 18 PET scan, CT scan, and ferumoxtran-10 MRI scan finds lymph node metastasis before undergoing chemotherapy and radiation therapy in patients with locally advanced cervical cancer or high-risk endometrial cancer. Diagnostic procedures, such as a fludeoxyglucose F 18 positron emission tomography (PET) scan, computed tomography (CT) scan, and ferumoxtran-10 magnetic resonance imaging (MRI) scan, may help find lymph node metastasis in patients with cervical cancer or endometrial cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the diagnostic sensitivity and specificity of preoperative fludeoxyglucose F 18 positron emission tomography (FDG-PET)/CT scanning and ferumoxtran-10 MRI scanning in identifying metastases to abdominal (common iliac, para-aortic, and paracaval) lymph nodes in patients with locoregionally advanced cervical carcinoma.

II. Determine the diagnostic sensitivity and specificity of preoperative FDG-PET/CT scanning and ferumoxtran-10 MRI scanning in identifying metastases to retroperitoneal abdominal lymph nodes in patients with high-risk endometrial cancer.

SECONDARY OBJECTIVES:

I. Determine the diagnostic sensitivity and specificity of preoperative FDG-PET/CT scanning and ferumoxtran-10 MRI scanning in identifying metastases to pelvic lymph nodes and pelvic and abdominal lymph nodes combined in patients with locoregionally advanced cervical carcinoma or high-risk endometrial cancer.

II. Compare the additive diagnostic value of CT fusion (PET/CT scan) vs PET scanning alone in identifying metastases to pelvic, abdominal, and combined (all regions) lymph nodes in these patients.

III. Compare the diagnostic sensitivity and specificity of PET/CT scanning vs ferumoxtran-10 MRI scanning in identifying metastases to pelvic, abdominal, and combined lymph nodes in these patients.

IV. Compare the diagnostic sensitivity and specificity of ferumoxtran-10 MRI vs MRI alone, in terms of size criteria in the abdomen and pelvis, in these patients.

V. Determine the percentage of patients with locoregionally advanced cervical cancer or high-risk endometrial cancer who have biopsy-proven disease outside the abdominal or pelvic lymph nodes detected by PET/CT scanning.

VI. Determine the accuracy of MRI in determining the depth of myometrial invasion and involvement of cervix in patients with high-risk endometrial cancer.

VII. Determine the complications associated with extraperitoneal or laparoscopic abdominal and pelvic lymphadenectomy in patients with locoregionally advanced cervical cancer.

VIII. Determine the cause(s) of delay in the initiation of radiotherapy or interruption in radiotherapy in patients with locoregionally advanced cervical cancer.

IX. Collect data on the adverse effects of ferumoxtran-10 in patients with locoregionally advanced cervical carcinoma or high-risk endometrial cancer.

X. Compare the size of lymph nodes in pre- and post-ferumoxtran-10 MRI's in a subset of forty patients.

OUTLINE: This is a multicenter study.

Patients receive fludeoxyglucose F 18 (FDG) IV followed 60 minutes later by positron emission tomography (PET)/CT scanning on day 1. Patients also receive ferumoxtran-10 IV over 30-45 minutes on day 1 (or 24-36 hours before MRI) and undergo MRI on day 2. Patients undergo extraperitoneal, laparoscopic, or trans-peritoneal lymphadenectomy with pelvic and abdominal lymph node biopsy within 2 weeks after PET/CT scan. Patients diagnosed with metastatic disease prior to lymph node biopsy proceed directly to primary treatment. Patients with cervical cancer undergo chemoradiotherapy within 4 weeks of PET/CT scan.

After completion of study therapy, patients are followed at 6 weeks, 6 months, every 3 months for 2 years, and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of 1 of the following:

  * Invasive carcinoma of the cervix meeting all of the following criteria:

    * Previously untreated, primary disease
    * Locoregionally advanced (stage IB2, IIA [>= 4 cm], or IIB-IVA) disease
    * Any cell type allowed
  * High-risk endometrial carcinoma meeting 1 of the following criteria:

    * Grade 3 endometrioid or non-endometrioid endometrial carcinoma (clear cell or serous papillary) or carcinosarcoma diagnosed from an endometrial biopsy or dilation and curettage or
    * Grade 1 or 2 endometrioid endometrial carcinoma with cervical stromal involvement overt on clinical examination or confirmed by endocervical curettage
* Under consideration for chemoradiotherapy (patients with cervical cancer)
* Undergone appropriate surgery for cervical or endometrial carcinoma with appropriate tissue available for histologic evaluation to confirm diagnosis and stage
* Appropriate surgical candidate to undergo extraperitoneal or laparoscopic lymph node sampling OR hysterectomy and lymph node sampling

  * No surgery for patients with advanced lymphadenopathy
* No recurrent invasive carcinoma of the uterus or uterine cervix regardless of previous treatment
* No known metastases to the lungs or scalene lymph nodes
* No metastases to other organs outside of the pelvis or abdominal lymph nodes at the time of the original clinical diagnosis

  * Patients with endometrial cancer with known intraperitoneal disease are eligible provided they undergo pelvic and para-aortic lymphadenectomy per protocol
* Participants must be enrolled at an American College of Radiology Imaging Network (ACRIN)-affiliated institution that is accredited by Gynecologic Oncology Group (GOG)
* GOG performance status 0-2
* Creatinine within normal institutional limits OR, in participants with creatinine levels above institutional normal, glomerular filtration rate (GFR) must be > 60 mL/min; there is no lower limit of normal for serum creatinine for this protocol
* Ferritin levels =< 600 ng/mL OR saturation of transferrin level =< 50%

  * Patients with high levels of ferritin or transferrin are eligible if documented hematology rules out iron overload
* Not pregnant or nursing
* Negative pregnancy test
* No patients weighing greater than that allowable by the PET/CT scanner
* No renal abnormalities, such as a pelvic kidney, horseshoe kidney, or renal transplantation, that would require modification of the lymphadenectomy
* No history of anaphylactic or life-threatening allergic reactions to any contrast media
* No other invasive malignancies within the past 5 years with the exception of nonmelanoma skin cancer
* No contraindication to MRI (e.g., severe claustrophobia, pacemaker, aneurysm clips, defibrillators, or other institutional contraindication to MRI)
* No history of allergic reactions attributed to compounds of similar chemical or biological composition to ferumoxtran-10 (e.g., iron preparations, parenteral iron, parenteral dextran, parenteral iron-dextran, or parenteral iron-polysaccharide preparations)
* No immunodeficiencies that would predispose patient to specific or nonspecific mediator release
* No history of cirrhosis
* No poorly controlled, insulin-dependent diabetes (i.e., fasting blood glucose level > 200 mg/dL)
* No prior pelvic or abdominal lymphadenectomy
* No prior pelvic radiotherapy
* No prior anticancer therapy that would contraindicate study participation
* No ferumoxides within the past 2 weeks
* No investigational agents within the past 30 days
* No other concurrent investigational agents

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 384 (Actual)
Dates: Start 2007-09; Primary Completion 2014-09 (Actual); Study Completion 2016-07-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa Atri, Principal Investigator — NRG Oncology
Locations (33):
- United States (24):
  - Jonsson Comprehensive Cancer Center, Los Angeles, California
  - University of California at Los Angeles Health System, Los Angeles, California
  - Olive View-University of California Los Angeles Medical Center, Sylmar, California
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Georgia Regents University Medical Center, Augusta, Georgia
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - UMDNJ - New Jersey Medical School, Newark, New Jersey
  - Island Gynecologic Oncology, Brightwaters, New York
  - Mount Sinai Medical Center, New York, New York
  - Weill Medical College of Cornell University, New York, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Providence Cancer Center -The Plaza, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Brooke Army Medical Center, Fort Sam Houston, Texas
- CHUQ - Pavilion Hotel-Dieu de Quebec, Québec, Quebec, Canada
- Japan (3):
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Kagoshima City Hospital, Kagoshima City, Kagoshima
  - Saitama Medical University International Medical Center, Saitama
- South Korea (5):
  - Keimyung University-Dongsan Medical Center, Jung-Ku, Daegu
  - Seoul National University Hospital, Seoul
  - Gangnam Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Korea Cancer Center Hospital, Seoul

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on 9/24/2007. Combidex MRI was discontinued on 11/09/2009 due to lack of study drug. GOG 0233 (NCT 00416455) closed to accrual on 6/21/2013.
Groups:
- Cervical Cancer Patients: PET/CT 60 minutes after FDG IV on day 1; Combidex IV over 30 - 45 minutes, day 1 (or 24-36 hours before MRI). MRI on day 2; Extraperitoneal, laparoscopic, or trans-peritoneal lymphadenectomy with pelvic and abdominal lymph node biopsy within 2 weeks after PET/CT scan
- Endometrial Cancer Patients: PET/CT 60 minutes after FDG IV on day 1; Extraperitoneal, laparoscopic, or trans-peritoneal lymphadenectomy with pelvic and abdominal lymph node biopsy within 2 weeks after PET/CT scan
Period: Overall Study
Arm/Group | Cervical Cancer Patients | Endometrial Cancer Patients
Started | 169 (This is a diagnostic imaging study.) | 215 (This is a diagnostic imaging study.)
Completed | 153 (Number of patients with adequate imaging and pathology) | 207 (Number of patients with adequate imaging and pathology)
Not Completed | 16 | 8
Not completed — PET / CT not done | 3 | 5
Not completed — PET / CT poor quality | 2 | 1
Not completed — Inadequate pathology | 11 | 2

BASELINE CHARACTERISTICS:
Population: Adequate imaging and pathologically eligible patients (N =360)
Groups:
- Total: Total of all reporting groups
Arm/Group | Cervical Cancer Patients | Endometrial Cancer Patients | Total
Number analyzed (Participants) | 153 | 207 | 360
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (11.6) | 64.8 (9.9) | 58 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 153 | 207 | 360
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Diagnostic Sensitivity of PET/CT for Detection of Lymph Node Metastasis in Abdomen
Description: The sensitivity is defined as the percentage of patients who test with lymph node metastases by pre-operative PET/CT among the patients who have lymph node metastases identified by post-surgery pathology in abdomen. The reported sensitivity is reader average sensitivity by seven experienced PET-CT readers.
Time Frame: Before surgery (FDG-PET-CT) and after surgery (pathology)
Population: Abdominal positive and negative patients. Cervix cohort, first 40 abdominal positive and 40 randomly selected abdominal negative patients. Endometrial cancer cohort, all 23 abdominal positive and 26 randomly selected abdominal negative patients
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cervical Cancer Patients | Endometrial Cancer Patients
Number analyzed (Participants) | 80 | 49
percentage of participants | 50 [44 to 56] | 65 [57 to 72]

2. Primary Outcome: The Diagnostic Specificity of PET/CT for Detection of Lymph Node Metastasis in Abdomen
Description: The specificity is defined as the percentage of patients who test without lymph node metastases by pre-operative PET/CT among the patients who do not have lymph node metastases identified by post-surgery pathology in abdomen. The reported specificity is reader average specificity by seven experienced PET-CT readers.
Time Frame: Before surgery (FDG-PET/CT) and after surgery (pathology)
Population: Patients with abdominal positive and negative lymph nodes. Cervix cohort, first 40 abdominal positive and 40 randomly selected abdominal negative patients. Endometrial cancer cohort, all 23 abdominal positive and 26 randomly selected abdominal negative patients.
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cervical Cancer Patients | Endometrial Cancer Patients
Number analyzed (Participants) | 80 | 49
percentage of participants | 85 [80 to 89] | 88 [83 to 92]

3. Secondary Outcome: The Diagnostic Sensitivity of PET/CT for Detection of Lymph Node Metastasis in Pelvis
Description: The sensitivity is defined as the percentage of patients who test with lymph node metastases by pre-operative PET/CT among the patients who have lymph node metastases identified by post-surgery pathology in pelvis. The reported sensitivity is reader-averaged sensitivity.
Time Frame: Before surgery (DCT) and after surgery (pathology)
Population: Patients with abdominal positive and negative lymph nodes. Cervical cancer cohort, first 40 abdominal positive and 40 randomly selected abdominal negative patients. Endometrial cancer cohort, all 23 abdominal positive and 26 randomly selected abdominal negative patients.
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cervical Cancer Patients | Endometrial Cancer Patients
Number analyzed (Participants) | 80 | 49
percentage of participants | 83 [78 to 87] | 65 [57 to 72]

4. Secondary Outcome: The Diagnostic Specificity of PET/CT for Detection of Lymph Node Metastasis in Pelvis
Description: The specificity is defined as the percentage of patients who test without lymph node metastases in pelvis by pre-operative PET/CT among the patients who do not have lymph node metastases in pelvis identified by post-surgery pathology. The reported specificity is reader-averaged specificity.
Time Frame: Before surgery (FDG-PET/CT) and after surgery (pathology)
Population: Cervix cohort, first 40 abdominal positive and 40 randomly selected abdominal negative patients. Endometrial cancer cohort, all 23 abdominal positive and 26 randomly selected abdominal negative patients
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cervical Cancer Patients | Endometrial Cancer Patients
Number analyzed (Participants) | 80 | 49
percentage of participants | 63 [54 to 70] | 93 [86 to 96]

5. Secondary Outcome: The Diagnostic Sensitivity of PET/CT for Detection of Lymph Node Metastasis in Combination of Abdomen and Pelvis
Description: The sensitivity is defined as the percentage of patients who test with lymph node metastases by pre-operative PET/CT among the patients who have lymph node metastases identified by post-surgery pathology in combination of abdomen and pelvis. The reported sensitivity is reader-average sensitivity.
Time Frame: Before surgery (FDG-PET/CT) and after surgery (pathology)
Population: Patients with abdominal positive and negative lymph nodes. Cervix cohort, first 40 abdominal positive and 40 randomly selected abdominal negative patients Endometrial cancer cohort, all 23 abdominal positive and 26 randomly selected abdominal negative patients
Measure: Mean (95% Confidence Interval); unit: Percentage of participants
Groups:
- Cervical Cancer Patients: PET/CT 60 minutes after FDG IV on day 1; Combidex IV over 30 - 45 minutes, day 1 (or 24-36 hours before MRI). MRI on day 2; Extraperitoneal, laparoscopic, or trans-peritoneal lymphadenectomy with pelvic and abdominal lymph node biopsy within 2 weeks after PET/CT scan. Cervix cohort, first 40 abdominal positive and 40 randomly selected abdominal negative patients.
- Endometrial Cancer Patients: PET/CT 60 minutes after FDG IV on day 1; Extraperitoneal, laparoscopic, or trans-peritoneal lymphadenectomy with pelvic and abdominal lymph node biopsy within 2 weeks after PET/CT scan. Endometrial cancer cohort, all 23 abdominal positive and 26 randomly selected abdominal negative patients
Arm/Group | Cervical Cancer Patients | Endometrial Cancer Patients
Number analyzed (Participants) | 80 | 49
Percentage of participants | 81 [77 to 85] | 63 [56 to 70]

6. Secondary Outcome: The Diagnostic Specificity of PET/CT for Detection of Lymph Node Metastasis in Combination of Abdomen and Pelvis
Description: The specificity is defined as the percentage of patients who test without lymph node metastases by pre-operative PET/CT among the patients who do not have lymph node metastases identified by post-surgery pathology in combination of abdomen and pelvis. The reported specificity is reader-averaged specificity.
Time Frame: Before surgery (FDG-PET/CT) and after surgery (pathology)
Population: Cervical cohort, first 40 abdominal positive and 40 randomly selected abdominal negative patients. Endometrial cancer cohort, all 23 abdominal positive and 26 randomly selected abdominal negative patients.
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cervical Cancer Patients | Endometrial Cancer Patients
Number analyzed (Participants) | 80 | 49
percentage of participants | 69 [59 to 77] | 83 [76 to 88]

7. Secondary Outcome: Sensitivity for Detection of Lymph Node Metastasis in Abdomen by CT Alone
Description: The sensitivity is defined as the percentage of patients who test with lymph node metastases by pre-operative CT alone among the patients who have lymph node metastases identified by post-surgery pathology in abdomen. The reported estimate of sensitivity is reader-average sensitivity across all 7 experienced PET-CT readers.
Time Frame: Before surgery (FDG-PET/CT) and after surgery (pathology)
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Groups:
- Cervical Cancer Patients - Sensitivity of CT: CT 60 minutes after FDG IV on day 1; Combidex IV over 30 - 45 minutes, day 1 (or 24-36 hours before MRI). MRI on day 2; Extraperitoneal, laparoscopic, or trans-peritoneal lymphadenectomy with pelvic and abdominal lymph node biopsy within 2 weeks after PET/CT scan. Cervix cohort, first 40 abdominal positive and 40 randomly selected abdominal negative patients.
- Endometrial Cancer Cohort - Sensitivity of CT: CT 60 minutes after FDG IV on day 1; Extraperitoneal, laparoscopic, or trans-peritoneal lymphadenectomy with pelvic and abdominal lymph node biopsy within 2 weeks after CT scan. Endometrial cancer cohort, all 23 abdominal positive and 26 randomly selected abdominal negative patients
Arm/Group | Cervical Cancer Patients - Sensitivity of CT | Endometrial Cancer Cohort - Sensitivity of CT
Number analyzed (Participants) | 80 | 49
percentage of participants | 42 [36 to 48] | 50 [43 to 58]

8. Secondary Outcome: Sensitivity for Detection of Lymph Node Metastasis in Pelvis by CT Alone
Description: The sensitivity is defined as the percentage of patients who test with lymph node metastases by pre-operative either CT alone among the patients who have lymph node metastases identified by post-surgery pathology in pelvis. The reported estimate of sensitivity is reader-average sensitivity across all 7 experienced PET-CT readers.
Time Frame: Before surgery (FDG-PET/CT) and after surgery (pathology)
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Groups:
- Cervical Cancer Patients - Sensitivity of CT: CT 60 minutes after FDG IV on day 1; Combidex IV over 30 - 45 minutes, day 1 (or 24-36 hours before MRI). MRI on day 2; Extraperitoneal, laparoscopic, or trans-peritoneal lymphadenectomy with pelvic and abdominal lymph node biopsy within 2 weeks after CT scan
- Endometrial Cancer Cohort - Sensitivity of CT: CT 60 minutes after FDG IV on day 1; Extraperitoneal, laparoscopic, or trans-peritoneal lymphadenectomy with pelvic and abdominal lymph node biopsy within 2 weeks after CT scan
Arm/Group | Cervical Cancer Patients - Sensitivity of CT | Endometrial Cancer Cohort - Sensitivity of CT
Number analyzed (Participants) | 80 | 49
percentage of participants | 79 [73 to 83] | 48 [41 to 56]

9. Secondary Outcome: Sensitivity Between for Detection of Lymph Node Metastasis in Combination of Abdomen and Pelvis by CT Alone
Description: The sensitivity is defined as the percentage of patients who test with lymph node metastases by pre-operative by CT alone among the patients who have lymph node metastases identified by post-surgery pathology in pelvis. The reported estimate of sensitivity is reader-average sensitivity across all 7 experienced PET-CT readers.
Time Frame: Before surgery (FDG-PET/CT) and after surgery (pathology)
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Groups:
- Cervical Cancer Patients-Sensitivity of CT: CT 60 minutes after FDG IV on day 1; Combidex IV over 30 - 45 minutes, day 1 (or 24-36 hours before MRI). MRI on day 2; Extraperitoneal, laparoscopic, or trans-peritoneal lymphadenectomy with pelvic and abdominal lymph node biopsy within 2 weeks after CT scan
- Endometrial Cancer Patients: CT 60 minutes after FDG IV on day 1; Extraperitoneal, laparoscopic, or trans-peritoneal lymphadenectomy with pelvic and abdominal lymph node biopsy within 2 weeks after PET/CT scan
Arm/Group | Cervical Cancer Patients-Sensitivity of CT | Endometrial Cancer Patients
Number analyzed (Participants) | 80 | 49
percentage of participants | 77 [73 to 81] | 54 [47 to 61]

10. Secondary Outcome: Specificity for Detection of Lymph Node Metastasis in Abdomen by CT Alone
Description: The specificity is defined as the percentage of patients who test without lymph node metastases by pre-operative CT alone among the patients who do not have lymph node metastases identified by post-surgery pathology in pelvis. The reported estimate of specificity is reader-average specificity across all 7 experienced PET-CT readers.
Time Frame: Before surgery (FDG-PET/CT) and after surgery (pathology)
Population: Patients with abdominal positive and negative lymph nodes. Cervical cancer cohort, first 40 abdominal positive and 40 randomly selected abdominal negative patients Endometrial cancer cohort, all 23 abdominal positive and 26 randomly selected abdominal negative patients
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cervical Cancer Patients | Endometrial Cancer Patients
Number analyzed (Participants) | 80 | 49
percentage of participants | 89 [84 to 92] | 93 [89 to 96]

11. Secondary Outcome: Specificity Between for Detection of Lymph Node Metastasis in Pelvis by CT Alone
Description: The specificity is defined as the percentage of patients who test without lymph node metastases by pre-operative byCT alone among the patients who do not have lymph node metastases identified by post-surgery pathology in pelvis. The reported estimate of specificity is reader-average specificity across all 7 experienced PET-CT readers.
Time Frame: Before surgery (FDG-PET/CT) and after surgery (pathology)
Population: Patients with abdominal positive and negative lymph nodes. Cervical cancer cohort, first 40 abdominal positive and 40 randomly selected abdominal negative patients. Endometrial cancer cohort, all 23 abdominal positive and 23 randomly selected abdominal negative patients
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cervical Cancer Patients | Endometrial Cancer Patients
Number analyzed (Participants) | 80 | 49
percentage of participants | 62 [53 to 69] | 89 [82 to 94]

12. Secondary Outcome: Specificity for Detection of Lymph Node Metastasis in Combination of Abdomen and Pelvis by CT Alone
Description: as for outcome 10
Time Frame: Before surgery (FDG-PET/CT) and after surgery (pathology)
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cervical Cancer Patients | Endometrial Cancer Patients
Number analyzed (Participants) | 80 | 49
percentage of participants | 63 [54 to 72] | 85 [78 to 90]

13. Secondary Outcome: Percentage of Participants in Whom PET/CT Detects Biopsy-proven Disease Outside the Abdominal Lymph Nodes
Time Frame: Before surgery (FDG-PET/CT) and after surgery (pathology)
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Cervical Cancer Patients | Endometrial Cancer Patients
Number analyzed (Participants) | 80 | 49
percentage of participants | 9 | 10

14. Secondary Outcome: Percentage of Participants in Whom PET/CT Detects Biopsy-proven Disease Outside the Pelvic Lymph Node
Time Frame: Before surgery (FDG-PET/CT) and after surgery (pathology)
Population: Particpants with abdominal positive and negative lymph nodes. Cervical cancer cohort, first 40 abdominal positive and 40 randomly selected abdominal negative patients. Endometrial cancer cohort, all 23 abdominal positive and 26 randomly selected abdominal negative patients
Measure: Number; unit: percentage of participants
Arm/Group | Cervical Cancer Patients | Endometrial Cancer Patients
Number analyzed (Participants) | 80 | 49
percentage of participants | 10 | 6

15. Secondary Outcome: Cervical Cancer Patients With Adverse Events (Grade 3 or Higher) at Least Possibly Attributed to Extra-peritoneal or Laparoscopic Abdominal and Pelvic Lymphadenectomy
Description: Number of participants with cervical cancer and a maximum grade of 3 or higher during treatment period. Adverse events are graded and categorized using CTCAE v3.0.
Time Frame: During surgery and up to 30 days after surgery.
Population: All loco-regionally advanced cervical cancer patients who had extra-peritoneal or laparoscopic abdominal and pelvic lymphadenectomy
Measure: Count of Participants; unit: Participants
Groups:
- Number of Participants With a Maximum Grade of 3 or Higher Dur: Number of participants with a maximum grade of 3 or higher during treatment period and up to 30 days after stopping study treatment.
Arm/Group | Number of Participants With a Maximum Grade of 3 or Higher Dur
Number analyzed (Participants) | 127
Participants
  Leukopenia | 1
  Thrombocytopenia | 1
  Anemia | 7
  Other Hematologic | 1
  Dermatologic | 1
  Gastrointestinal | 4
  Infection | 9
  Lymphatics | 5
  Metabolic | 3
  Musculoskeletal | 1
  Pain | 2
  Vascular | 3

16. Secondary Outcome: Cause of Delay in the Initiation of Chemo-radiation Therapy More Than 4 Weeks After PET/CT for Cervical Cancer Patients
Description: Number of cervical cancer patients with reasons of delay in the initiation of chemo-radiation therapy
Time Frame: Within 4 weeks from PET/CT
Population: All Loco-regionally advanced cervical cancer patients who had extra-peritoneal or laparoscopic abdominal and pelvic lymphadenectomy and the reason they experienced a delay in the initiation of chemo-radiation
Measure: Count of Participants; unit: Participants
Groups:
- Cause of Delay in the Initiation of Chemo-radiation Therapy mo: All Loco-regionally advanced cervical cancer patients who had extra-peritoneal or laparoscopic abdominal and pelvic lymphadenectomy who experienced a delay in the initiation of chemo-radiation therapy
Arm/Group | Cause of Delay in the Initiation of Chemo-radiation Therapy mo
Number analyzed (Participants) | 127
Participants
  Surgery related adverse events | 3
  Patient preference/scheduling difficulty | 21
  Other | 6
  Not reported | 3
  No Delay | 94

17. Secondary Outcome: Cause of Interruption in Radiation Therapy in Cervical Cancer Patients
Description: Number of cervical cancer patients with reasons of interruption in radiation therapy
Time Frame: Within 6 weeks after surgery
Population: Loco-regionally advanced cervical cancer patients who had extra-peritoneal or laparoscopic abdominal and pelvic lymphadenectomy who experienced an interruption in radiation therapy
Measure: Count of Participants; unit: Participants
Groups:
- Causes of Interruption in Radiation Therapy: Number of participants with reasons of interruption in radiation therapy
Arm/Group | Causes of Interruption in Radiation Therapy
Number analyzed (Participants) | 127
Participants
  Chemoradiation related adverse events | 1
  Patient preference/scheduling difficulty | 1
  Other | 9
  Not reported | 14
  No interruption | 102

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) occurring within 30 days of surgery are reported
Arm/Group | Cervical Cancer Patients | Endometrial Cancer Patients
Serious Adverse Events (participants affected / at risk) | 17/169 | 19/215
Other Adverse Events (participants affected / at risk) | 108/169 | 132/215
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cervical Cancer Patients (N=169) | Endometrial Cancer Patients (N=215)
Conduction Abnml: Asystole (Cardiac disorders) | 0 | 1
S/N Arrhythmia: Atrial Flutter (Cardiac disorders) | 0 | 1
Hypotension (Cardiac disorders) | 1 | 0
Death No Ctcae Term - Death Nos (General disorders) | 0 | 1
Fistula, Gi - Colon/Cecum/Appendix (Gastrointestinal disorders) | 1 | 0
Obstruction, Gi - Colon (Gastrointestinal disorders) | 1 | 0
Obstruction, Gi - Small Bowel Nos (Gastrointestinal disorders) | 0 | 3
Dehydration (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Hemorrhage, Gu - Vagina (Vascular disorders) | 0 | 1
Hemorrhage With Surgery (Vascular disorders) | 0 | 1
Hemorrhage, Gi - Abdomen Nos (Vascular disorders) | 0 | 1
Hemorrhage/Bleeding - Other (Vascular disorders) | 1 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Wound (Infections and infestations) | 2 | 0
Inf Unknown Anc: Lung (Pneumonia) (Infections and infestations) | 0 | 1
Infection - Other (Infections and infestations) | 1 | 0
Inf Unknown Anc: Pelvis Nos (Infections and infestations) | 1 | 1
Inf Unknown Anc: Lymphatic (Infections and infestations) | 1 | 0
Inf Unknown Anc: Small Bowel Nos (Infections and infestations) | 0 | 1
Inf Unknown Anc: Abdomen Nos (Infections and infestations) | 0 | 1
Inf Unknown Anc: Skin (Cellulitis) (Infections and infestations) | 1 | 0
Lymphocele (Blood and lymphatic system disorders) | 0 | 1
Pain: Gallbladder (General disorders) | 1 | 0
Pain: Abdominal Pain Nos (General disorders) | 1 | 0
Leak, Gu - Ureter (Renal and urinary disorders) | 0 | 1
2nd Mal: Poss. Related To Cancer Rx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Intra-Op Injury: Other (Surgical and medical procedures) | 0 | 1
Tumor Flare (General disorders) | 1 | 0
Thrombosis/Embolism (Vascular Access-Related) (Vascular disorders) | 1 | 0
Thrombosis/Thrombus/Embolism (Vascular disorders) | 2 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cervical Cancer Patients (N=169) | Endometrial Cancer Patients (N=215)
Neutrophils (Blood and lymphatic system disorders) | 6 | 6
Platelets (Blood and lymphatic system disorders) | 19 | 11
Blood/Bone Marrow - Other (Blood and lymphatic system disorders) | 3 | 3
Leukocytes (Blood and lymphatic system disorders) | 24 | 13
Lymphopenia (Blood and lymphatic system disorders) | 2 | 2
Hemoglobin (Blood and lymphatic system disorders) | 80 | 88
S/N Arrhythmia: Atrial Fibrillation (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 1 | 1
Conduction Abnml: Asystole (Cardiac disorders) | 0 | 1
S/N Arrhythmia: Atrial Flutter (Cardiac disorders) | 0 | 1
S/N Arrhythmia: Sinus Tachycardia (Cardiac disorders) | 1 | 1
S/N Arrhythmia: Sinus Bradycardia (Cardiac disorders) | 0 | 1
Hypertension (Cardiac disorders) | 0 | 1
Hypotension (Cardiac disorders) | 3 | 2
Inr (Vascular disorders) | 0 | 2
Coagulopathy - Other (Vascular disorders) | 1 | 0
Weight Gain (General disorders) | 1 | 0
Fever (General disorders) | 6 | 4
Weight Loss (General disorders) | 2 | 1
Rigors/Chills (General disorders) | 2 | 0
Fatigue (General disorders) | 7 | 11
Insomnia (General disorders) | 0 | 1
Death No Ctcae Term - Disease Progression Nos (General disorders) | 1 | 0
Death No Ctcae Term - Death Nos (General disorders) | 0 | 1
Hair Loss/Alopecia (Scalp Or Body) (Skin and subcutaneous tissue disorders) | 0 | 1
Wound Complication, Non-Infectious (Skin and subcutaneous tissue disorders) | 1 | 7
Bruising (Skin and subcutaneous tissue disorders) | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 3 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 2 | 0
Hot Flashes (Endocrine disorders) | 0 | 1
Fistula, Gi - Colon/Cecum/Appendix (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 3 | 1
Hemorrhoids (Gastrointestinal disorders) | 0 | 1
Heartburn (Gastrointestinal disorders) | 1 | 0
Leak, Gi - Leak Nos (Gastrointestinal disorders) | 0 | 1
Fistula, Gi - Jejunum (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 2 | 7
Distention (Gastrointestinal disorders) | 1 | 0
Dry Mouth (Gastrointestinal disorders) | 1 | 0
Obstruction, Gi - Small Bowel Nos (Gastrointestinal disorders) | 2 | 2
Colitis (Gastrointestinal disorders) | 1 | 0
Obstruction, Gi - Jejunum (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 8 | 7
Anorexia (Gastrointestinal disorders) | 9 | 8
Dehydration (Gastrointestinal disorders) | 3 | 2
Constipation (Gastrointestinal disorders) | 12 | 10
Nausea (Gastrointestinal disorders) | 18 | 12
Gastrointestinal - Other (Gastrointestinal disorders) | 0 | 2
Diarrhea (Gastrointestinal disorders) | 6 | 4
Hemorrhage, Gu - Vagina (Vascular disorders) | 6 | 2
Hemorrhage, Gi - Upper Gi Nos (Vascular disorders) | 1 | 0
Hematoma (Vascular disorders) | 0 | 2
Hemorrhage, Gi - Abdomen Nos (Vascular disorders) | 0 | 1
Petechiae (Vascular disorders) | 1 | 0
Hemorrhage/Bleeding - Other (Vascular disorders) | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Lung(Pneumonia) (Infections and infestations) | 0 | 3
Inf W/Nml Or Gr 1 Or 2 Anc: Wound (Infections and infestations) | 3 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Skin(Cellulitis) (Infections and infestations) | 1 | 0
Inf Unknown Anc: Lung (Pneumonia) (Infections and infestations) | 0 | 2
Inf W/Nml Or Gr 1 Or 2 Anc: Colon (Infections and infestations) | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Urinary Tract Nos (Infections and infestations) | 4 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Abdomen Nos (Infections and infestations) | 1 | 0
Infection - Other (Infections and infestations) | 0 | 1
Colitis, Infectious (Eg.C. Difficile) (Infections and infestations) | 1 | 1
Inf Unknown Anc: Pelvis Nos (Infections and infestations) | 1 | 1
Inf Unknown Anc: Upper Airway Nos (Infections and infestations) | 1 | 0
Inf Unknown Anc: Bronchus (Infections and infestations) | 0 | 1
Inf Unknown Anc: Urinary Tract Nos (Infections and infestations) | 2 | 3
Inf Unknown Anc: Wound (Infections and infestations) | 1 | 1
Inf Unknown Anc: Abdomen Nos (Infections and infestations) | 0 | 1
Inf Unknown Anc: Skin (Cellulitis) (Infections and infestations) | 1 | 2
Inf W/Nml Or Gr 1 Or 2 Anc: Bladder (Infections and infestations) | 0 | 1
Lymphatics - Other (Blood and lymphatic system disorders) | 1 | 0
Lymphocele (Blood and lymphatic system disorders) | 6 | 1
Edema: Viscera (Blood and lymphatic system disorders) | 1 | 0
Edema: Trunk/Genital (Blood and lymphatic system disorders) | 2 | 0
Edema: Limb (Blood and lymphatic system disorders) | 3 | 5
Chyle Or Lymph Leakage (Blood and lymphatic system disorders) | 0 | 2
Ast (Metabolism and nutrition disorders) | 1 | 3
Metabolic/Laboratory - Other (Metabolism and nutrition disorders) | 2 | 1
Proteinuria (Metabolism and nutrition disorders) | 0 | 1
Hemoglobinuria (Metabolism and nutrition disorders) | 0 | 1
Creatinine (Metabolism and nutrition disorders) | 2 | 9
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 | 19
Alt (Metabolism and nutrition disorders) | 3 | 4
Alkaline Phosphatase (Metabolism and nutrition disorders) | 1 | 7
Hypermagnesemia (Metabolism and nutrition disorders) | 2 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 7
Hyponatremia (Metabolism and nutrition disorders) | 7 | 18
Hypernatremia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 15 | 52
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 5
Hyperglycemia (Metabolism and nutrition disorders) | 14 | 51
Hypokalemia (Metabolism and nutrition disorders) | 9 | 27
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 4 | 9
Musculoskeletal/St: Other (Musculoskeletal and connective tissue disorders) | 0 | 1
Soft Tissue Necrosis - Abdomen (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle Weakness - Whole Body/Generalized (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle Weakness - Extremity-Lower (Musculoskeletal and connective tissue disorders) | 1 | 0
Mental Status (Nervous system disorders) | 0 | 1
Mood Alteration - Depression (Nervous system disorders) | 1 | 0
Mood Alteration - Anxiety (Nervous system disorders) | 3 | 2
Dizziness (Nervous system disorders) | 2 | 0
Neuropathy-Sensory (Nervous system disorders) | 2 | 3
Neuropathy-Motor (Nervous system disorders) | 0 | 1
Pain - Other (General disorders) | 3 | 3
Pain: Urethra (General disorders) | 2 | 0
Pain: Pelvis (General disorders) | 5 | 0
Pain: Breast (General disorders) | 1 | 0
Pain: Vagina (General disorders) | 1 | 0
Pain: Chest /Thorax Nos (General disorders) | 1 | 1
Pain: Chest Wall (General disorders) | 0 | 1
Pain: Head/Headache (General disorders) | 4 | 0
Pain: Extremity-Limb (General disorders) | 4 | 2
Pain: Back (General disorders) | 4 | 2
Pain: Joint (General disorders) | 0 | 1
Pain: Gallbladder (General disorders) | 1 | 0
Pain: Abdominal Pain Nos (General disorders) | 12 | 14
Pain: Skin (General disorders) | 1 | 0
Pain: Muscle (General disorders) | 0 | 1
Pain: Anus (General disorders) | 1 | 0
Edema, Larynx (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Renal/Genitourinary - Other (Renal and urinary disorders) | 2 | 2
Leak, Gu - Ureter (Renal and urinary disorders) | 0 | 1
Cystitis (Renal and urinary disorders) | 1 | 0
Urinary Retention (Renal and urinary disorders) | 3 | 2
Obstruction, Gu - Ureter (Renal and urinary disorders) | 2 | 0
Incontinence, Urinary (Renal and urinary disorders) | 0 | 1
Bladder Spasm (Renal and urinary disorders) | 0 | 2
Renal Failure (Renal and urinary disorders) | 0 | 1
Urinary Frequency (Renal and urinary disorders) | 3 | 2
Vaginal Discharge (Reproductive system and breast disorders) | 2 | 1
Intra-Op Injury: Vein-Inferior Vena Cava (Surgical and medical procedures) | 0 | 1
Intra-Op Injury: Bladder (Surgical and medical procedures) | 0 | 1
Flu-Like Syndrome (General disorders) | 0 | 1
Thrombosis/Embolism (Vascular Access-Related) (Vascular disorders) | 1 | 2
Thrombosis/Thrombus/Embolism (Vascular disorders) | 4 | 1

LIMITATIONS AND CAVEATS:
Relatively small number of patients with abdominal metastasis in both cervical and endometrial cancer cohorts

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less